CLINICAL TRIAL: NCT05173467
Title: Robot-assisted Invasion-controlled Surgery Versus Traditional-open Surgery Against Metastatic Spinal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Wei Xu, Clinical Professor, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021SL046
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Minimally Invasive Surgery; Spinal Metastases
Keywords: Minimal surgery; Spinal Metastases; invsasion-controlled surgery; traditional-open surgery; Robot-assisted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted Invasion-controlled Surgery (Experimental)
  Interventions: Procedure: Robot-assisted Invasion-controlled Surgery
- Traditional-open Surgery (Placebo Comparator)
  Interventions: Procedure: Traditional-open Surgery

INTERVENTIONS:
Procedure: Robot-assisted Invasion-controlled Surgery — The concept of invasion-controlled surgery (ICS) for spinal metastasis has been put forward against the spinal instability and neurological dysfunction of frail patients that might not allowed for radical traditional open surgery including improvements of multidisciplinary dynamic assessments, endovascular detachable balloon embolization, minimal-invasion by using expandable working tubes, percutaneous pedicle screws, and some accurate therapy. ICS could provide immediate stability, deformity correction, and recovery of neurological function.
  Arms: Robot-assisted Invasion-controlled Surgery
Procedure: Traditional-open Surgery — This traditionally requires a midline incision, bilateral muscle strip, and multilevel laminectomy to provide adequate access and safe removal of the tumor.
  Arms: Traditional-open Surgery

SUMMARY:
With significant advances in diagnostic imaging and systemic therapies for oncologic disease, spinal metastasis with neurological dysfunction and mechanical instability has become an indication for surgery. Even if traditional-open surgery was palliative, the treatment of spinal metastasis also carried significant surgical morbidity. Those high morbidity and complication rates may influence the quality of patients with a limited life expectancy. Invasion-controlled surgery was utilized with Robot-assisted surgery approach against symptomatic spinal metastasis.

Increasing interest in the potential for improved consistency, complication reduction, and decreased length of hospitalization through robot utilization is evident from the rapid growth of publications seen in recent years.

So, the investigators wish to evaluate the advantages of Robot-assisted Invasion-controlled Surgery compared with traditional-open surgery spinal surgery in patients with metastatic spinal cord compression.

DETAILED DESCRIPTION:
Surgical Spinal Decompression of Metastatic Spinal Cord Compression, Minimal Access Versus Open Surgery. A prospective Clinical Trial

Purpose To investigate the effect of Robot-assisted Invasion-controlled Surgery compared with traditional-open surgery in the treatment of patients with metastatic spinalcord compression.

Hypotheses The group of patient's receiving robot-assisted invasion-controlled surgery will have better improvement in quality after surgery compared to the group that will receive traditional open surgery. The robot-assisted invasion-controlled surgery group will have reduction in per-operative bleeding and less wound complications compered to the group of patients receiving open or traditional surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of spinal metastasis (previously confirmed diagnosis of lung cancer, liver cancer, prostate cancer, breast cancer, kidney cancer, digestive tract cancer, imaging indicated the presence of metastatic lesions in the spine)
2. Patients with symptoms of spinal instability or nerve compression (SINS score of spinal instability ≥7, spinal nerve compression according to spinal cord injury Classification, grade A-D)
3. Metastases are located in the thoracic and/or lumbar vertebrae
4. The patient's expected survival was longer than 6 months
5. The subjects or their legal representatives were able to understand the study purpose, demonstrate adequate compliance with the study protocol, and sign informed consent

Exclusion Criteria:

1. He had previously operated on the same site
2. Spontaneous multiple compression fractures of the spine;
3. There is malformed osteitis (Paget's bone disease), osteomalacia, or other metabolic bone disease;
4. here were developmental vertebral malformations or vertebral body and pedicle dysplasia in the spinal segment to be treated by surgery
5. Presence of heart, lung, liver or kidney failure or other serious diseases (such as osteomyelitis, systemic infection, severe hemorrhagic disease, active disseminated intravascular coagulation, serious cardiovascular disease or myocardial infarction within 6 months prior to enrollment, cerebral infarction within 6 months prior to enrollment, severe psychiatric history)
6. Pregnant or lactating women
7. Participated in clinical trials of other drugs or medical devices within 3 months prior to enrollment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-25 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
operative bleeding | Intraoperative
  It is amount of blood lost during surgery, which is checked by the anesthesiologist and the surgical nurse.

SECONDARY OUTCOMES:
operation time | Intraoperative
  Is the time from the beginning of the operation to the end of the incision suture is the total operation time
Intraoperative transfusion volume | Intraoperative
  That is the amount of intraoperative red blood cell suspension and plasma input and the incidence of blood transfusion.
Intraoperative fluoroscopy dose | Intraoperative
  The product of intraoperative c-arm fluoroscopy times and single fluoroscopy dose
VAS Scores | less than 2 years
  It isrecorded at1D-3D after surgery (morning, middle and evening assessment every day, in which the most pain of each day was recorded. All patients were standardized to use the same dose of non-steroidal antipyretic and analgesic drugs; if temporary addition of A tablet analgesics was needed, VAS score before use was recorded and the dosage of A tablet was recorded), 2W after surgery, And 3M (long-term postoperative pain)
Frankel Scores | less than 2 years
  The Frankel Scale for Spinal Cord Injury That Classifies the Extent of the Neurological/Functional Deficit into Five Grades
Creatine kinase levels | less than 2 years
  reatine kinase were examined 1 day after operation
myoglobin | less than 2 years
  myoglobin were examined 1 day after operation
Complications | less than 2 years
  Postoperative wound complications were observed during the hospital period, including the incidence of wound infection, wound nonunion, wound debridement, and the frequency of massive bleeding, lung infection, urinary tract infection and other complications
QOL Scores | less than 2 years
  Quality of life (QOL) is a multidimensional concept that measures a person's wellbeing.
resuming time of daily life | less than 2 years
  Time spent in bed after surgery was recorded
Survival time | less than 2 years
  Survival time
ODI scores | less than 2 years
  The ODI is comprised of 10 questions. The questionnaire asks patients about their ability to manage everyday life and covers intensity of pain, lifting, the ability to care for oneself, ability to walk, the ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Answers are then scored on a 0-5 scale, zero meaning no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jianru Xiao, Profession, Study Chair — Shanghai Changzheng Hospital; Wei Xu, Profession, Study Director — Shanghai Changzheng Hospital; Bo Li, Profession, Principal Investigator — Shanghai Changzheng Hospital; Pengru Wang, Profession, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- ChangZheng Hospital, Shanghai, Shanghai Municipality, China